CLINICAL TRIAL: NCT05035680
Title: Proof of Concept Trial of Adjuvant Activity of SWE, a Squalene-based -Oil-in-water Emulsion
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study cancelled
Sponsor: Gates Medical Research Institute (Other)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MRI- ADV02-101
Record Dates: First submitted 2021-08-31; First posted 2021-09-05 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Influenza
Keywords: vaccine; influenza; adjuvant
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm i - Seasonal influenza vaccine (Active Comparator): Single 0.5 mL intramuscular (IM) injection of an unadjuvanted seasonal influenza vaccine
  Interventions: Biological: Unadjuvanted seasonal influenza vaccine
- Arm ii - SWE and unadjuvanted seasonal influenza vaccine (Experimental): Single 0.8 mL IM injection of SWE mixed with unadjuvanted seasonal influenza vaccine
  Interventions: Biological: SWE adjuvant mixed with unadjuvanted seasonal influenza vaccine shortly before dosing (SWE + QIV)
- Arm iii - MF59 adjuvanted seasonal influenza vaccine (Active Comparator): Single 0.5 mL IM injection of MF59 adjuvanted seasonal influenza vaccine
  Interventions: Biological: MF59 adjuvanted seasonal influenza vaccine

INTERVENTIONS:
Biological: Unadjuvanted seasonal influenza vaccine — Single 0.5 mL IM injection
  Arms: Arm i - Seasonal influenza vaccine
Biological: SWE adjuvant mixed with unadjuvanted seasonal influenza vaccine shortly before dosing (SWE + QIV) — Single 0.8 mL IM injection
  Arms: Arm ii - SWE and unadjuvanted seasonal influenza vaccine
Biological: MF59 adjuvanted seasonal influenza vaccine — Single 0.5 mL IM injection of MF59 adjuvanted seasonal influenza vaccine
  Arms: Arm iii - MF59 adjuvanted seasonal influenza vaccine

SUMMARY:
The purpose of the study is to characterize safety and tolerability of the squalene-based adjuvant candidate SWE and its potential to enhance the immune response to seasonal influenza vaccine antigens in healthy older adults.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing to participate in the study, as demonstrated by signing the written informed consent form approved by the Ethics Committee/Institutional Review Board (EC/IRB) before any study procedure is performed.
2. Be able to comprehend the full nature and purpose of the study, including possible risks.
3. Be a healthy male or female without acute or chronic medical condition per the Investigator's judgement between 18 to 50 years of age (Part 1) and ≥65 years of age (Part 2) on the day of randomization, inclusive.
4. Have a BMI between 18.0 kg/m2 and 32.0 kg/m2. BMI values should be rounded to the nearest integer (e.g., round down 32.4 to 32.0, round up 18.6 to 19.0).
5. All female participants: have a negative pregnancy test or post-menopausal status. Postmenopausal status is defined as 12 months with no menses without alternative medical cause. Female participants of childbearing potential (Part 1): have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day 1 prior to randomization, not breastfeeding, and willing to use highly effective methods of contraception 14 days before study drug administration through last scheduled follow up visit (End of Study). Male participants with female partners of child-bearing potential (Part 1): agree to use one of the following contraception methods from the day of randomization to the last follow-up visit of the partner: vasectomy with documentation of azoospermia, or male condom use; agree to not donate sperm prior to the last scheduled follow-up visit (End of Study).
6. Be able to co-operate with the study staff and comply with the requirements of the study.

Exclusion Criteria:

1. Have a history of intolerance, hypersensitivity, or allergy to any component of the study products and/or have a history of anaphylaxis to any drug or vaccines.
2. Have a history of Guillain-Barre Syndrome
3. Have a clinically significant history of hepatic, renal, cardiovascular, or any other disease or disorder, including psychological or psychiatric, that in the investigator's opinion may increase the risk to the participant, and/or jeopardize the participant's compliance with the study procedures.
4. Have a history of primary immunodeficiency or secondary immunodeficiency including HIV and anatomical or functional asplenia.
5. Have one or more abnormal laboratory values at the screening visit that in the opinion of the Investigator, are clinically significant, including but not limited to the following: Alanine Aminotransferase (ALT) > 2 x upper limit of normal (ULN) Serum creatinine above the ULN Bilirubin > 2 x ULN Internal Normalized Ratio (INR), Prothrombin Time (PT), Partial Thromboplastin Time (PTT) above the ULN Hemoglobin < 12 g/dL in men, and <11 g/dL in women Platelets below the lower limit of normal (LLN)
6. Have had clinical signs and symptoms consistent with Coronavirus Disease caused by severe acute respiratory syndrome coronavirus-2 (SARS-CoV2) infection-19 (COVID-19), i.e. fever, cough, dyspnea, sore throat, fatigue, loss of smell, loss of taste, or confirmed SARS-CoV-2 infection by appropriate laboratory test in the 1 month preceding the screening visit.
7. Have had influenza-like illness (ILI) in the 3 months preceding the screening visit. ILI is defined as fever (oral temperature ≥37.8 C / ≥100 F) and cough or sore throat (CDC definition).
8. Have received an investigational drug or vaccine in the 3 months preceding the screening visit, including COVID-19 investigational vaccine or treatment. Note: vaccination with an approved vaccine for the prevention of COVID-19 is allowed.
9. Have taken immunosuppressants and oral or parenteral corticosteroids in the 6 months preceding the screening visit. Inhaled corticosteroids for asthma are allowed.
10. Have received any influenza vaccine in the current and past season, i.e. in the 8 months preceding the screening visit.
11. Have a history of drug or alcohol abuse in the 1 year preceding the screening visit.
12. Have a history of basal cell carcinoma or non-invasive squamous cell carcinoma of the skin in the 1 year preceding the screening visit and/or a history of any other malignancy in the 5 years preceding the screening visit.
13. Have any other condition or situation that in the investigator's opinion might increase the risk to the participant or jeopardize the participant's compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-14 (Estimated); Primary Completion 2023-03-25 (Estimated); Study Completion 2023-11-25 (Estimated)

PRIMARY OUTCOMES:
Characterize the severe/serious adverse event (SAE) burden of SWE combined with a seasonal influenza vaccine over 28 days. | 7 days
  Severe systemic solicited AEs from Day 1 through Day 7
Characterize the severe/serious adverse event (SAE) burden of SWE combined with a seasonal influenza vaccine over 28 days. | 28 days
  Severe and serious unsolicited TEAEs from Day 1 through Day 28
Characterize the adjuvant effect of SWE on the hemagglutinin inhibition (HI) antibody response to the A/H3N2 vaccine strain. | Day 29
  HI antibody titer to the influenza A H3N2 (A/H3N2) vaccine strain on Day 29

SECONDARY OUTCOMES:
Characterize reactogenicity of SWE and MF59 combined with a seasonal influenza vaccine. | 7 days
  Local solicited AEs from Day 1 through Day 7
Characterize reactogenicity of SWE and MF59 combined with a seasonal influenza vaccine. | 7 days
  Systemic solicited AEs from Day 1 through Day 7
Characterize treatment-emergent adverse events (TEAEs) of SWE and MF59 combined with a seasonal influenza vaccine. | 28 Days
  TEAEs from Day 1 through Day 28
Characterize treatment-emergent adverse events (TEAEs) of SWE and MF59 combined with a seasonal influenza vaccine. | 169 Days (End of Study)
  SAEs from Day 1 through Day 169 (end of study)
Characterize safety laboratory values. | 29 Days and 169 Days (End of Study)
  Hematology assessments (complete blood count (red blood cells, hemoglobin, platelets and white blood cells) and differential (absolute counts) including neutrophils, lymphocytes, monocytes, eosinophils and basophils)) at 29 Days and 169 Days (End of Study)
Characterize safety laboratory values. | 29 Days and 169 Days (End of Study)
  Serum Chemistry assessments (ALT, AST, ALP, total bilirubin, creatinine, BUN, CRP, sodium and potassium, and chloride) at 29 Days and 169 Days (End of Study)
Characterize safety laboratory values. | 29 Days and 169 Days (End of Study)
  Serum Coagulation assessments (PT,PTT, and INR) at 29 Days and 169 Days (End of Study)
Characterize the adjuvant effect of SWE on HI antibody responses to homologous and heterologous influenza vaccine strains through HI antibody titer, peripheral blood mononuclear cell(PBMC), and exploratory laboratory assessments. | Day 29 and Day 169
  HI antibody titers to the homologous strains included in the vaccines on Day 29 and Day 169
Characterize the adjuvant effect of SWE on HI antibody responses to homologous and heterologous influenza vaccine strains through HI antibody titer, peripheral blood mononuclear cell(PBMC), and exploratory laboratory assessments. | Day 29 and Day 169
  HI antibody titers to the selected non vaccine (heterologous) strains on Day 29 and Day 169

CONTACTS AND LOCATIONS:
Overall Officials: BM Gates MRI, Study Chair — Gates Medical Research Institute

REFERENCES:
- See also: Fluad® Package Insert, 2021. — https://www.fda.gov/media/135432/download